CLINICAL TRIAL: NCT04812236
Title: A Randomized, Partially Double-blind, Controlled, Multi-center Clinical Study of Wulingsan Single Decoction Granules Combined With Conventional Therapy in the Treatment of Metabolic Syndrome of Spleen Deficiency, Dampness and Sleepiness
Brief Title: Clinical Study on Wuling Powder in Treating Metabolic Syndrome of Spleen Deficiency and Dampness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FM-P8-2018052801
Record Dates: First submitted 2021-02-22; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single decoction group: Wulingsan single decoction granules (Experimental): Wulingsan single decoction granules, Alisma orientalis (15g), Polyporus (10g), Baizhu (10g), Poria (10g), Guizhi (6g). Take 1 bag each time with warm water twice a day.Take 12 weeks as a course of treatment.
  Interventions: Drug: Wulingsan single decoction granules
- Co-decocting group: Wulingsan co-decocting granules (Other): Wulingsan co-decoction granules, Alisma orientalis (15g), Polyporus (10g), Atractylodes (10g), Poria (10g), Guizhi (6g). Take 1 bag each time with warm water twice a day.Take 12 weeks as a course of treatment.
  Interventions: Drug: Wulingsan co-decoction granules
- Powder group: Wuling powder powder (Other): Wuling powder is composed of Alisma, Polyporus, Atractylodes, Poria, Guizhi. Take 5g each time with warm water twice a day.Take 12 weeks as a course of treatment.
  Interventions: Drug: Wuling Powder
- Simulant group: Simulant of granular dosage form (Placebo Comparator): Granule simulant, the composition is Alisma orientalis (15g), Polyporus (10g), Atractylodes (10g), Poria (10g), Guizhi (6g). Take 1 bag each time with warm water twice a day. Take 12 weeks as a course of treatment.
  Interventions: Drug: Wulingsan granule simulant

INTERVENTIONS:
Drug: Wulingsan single decoction granules — Wulingsan single decoction granules, the prescription is Alisma, Polyporus, Atractylodes, Poria, Guizhi. Oral, 2 times a day, 2 sachets each time, rinsed with warm water
  Arms: Single decoction group: Wulingsan single decoction granules
Drug: Wulingsan co-decoction granules — Wulingsan co-decoction granules, the prescription is Alisma, Polyporus, Atractylodes, Poria, Guizhi. Oral, 2 times a day, 2 sachets each time, rinsed with warm water
  Arms: Co-decocting group: Wulingsan co-decocting granules
Drug: Wuling Powder — Wuling powder is composed of Alisma, Polyporus, Atractylodes, Poria, Guizhi. 2 times a day, 5g each time, take it with warm water
  Arms: Powder group: Wuling powder powder
Drug: Wulingsan granule simulant — Wulingsan granule simulant, the prescription is Alisma, Polyporus, Atractylodes, Poria, Guizhi. Oral, 2 times a day, 2 sachets each time, rinsed with warm water
  Arms: Simulant group: Simulant of granular dosage form

SUMMARY:
In this study, a randomized, partially double-blind, controlled, multi-center clinical research method was used. A total of 4 groups were designed, namely, single decoction group, co-decoction group, powder group and simulation group. The four groups of patients all received basic health education, diet control and increased exercise guidance. All the patients in the group have taken western medicine according to their own conditions and followed the doctor's instructions for hypoglycemic, blood pressure, and lipid-lowering treatments. After joining the group, they continue to take the medicine at the original dose, and the patients are advised not to change the medicine during the observation period. Take 12 weeks as a course of treatment, and set the observation period to 12 weeks. Follow up every 4 weeks.

DETAILED DESCRIPTION:
The research purpose of this project is to observe the effectiveness and safety of Wulingsan single decoction granules compared with traditional powder, co-decoction granules and analogues in the treatment of metabolic syndrome in combination with conventional therapies. ; Compared with Wulingsan traditional powder and co-decoction granule group, observe the effectiveness and safety of traditional powder combined with conventional therapy in the treatment of metabolic syndrome. The trial adopts a randomized, partially double-blind, controlled, multi-center clinical research method. A total of 320 cases were included in 4 groups, namely, single decoction group, co-decoction group, powder group, and simulated agent group. The four groups of patients all received basic health education, diet control and increased exercise guidance. All the patients in the group have taken western medicine according to their own conditions and followed the doctor's instructions for hypoglycemic, blood pressure, and lipid-lowering treatments. After joining the group, they continue to take the medicine at the original dose, and the patients are advised not to change the medicine during the observation period. Take 12 weeks as a course of treatment, and the observation period is set to 12 weeks. Follow up every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria of metabolic syndrome;
2. TCM syndrome differentiation of spleen deficiency and dampness patients;
3. Patients with phlegm-dampness constitution score>30;
4. Patients aged 18 to 70 years;
5. Patients who have signed informed consent and are highly compliant.

Exclusion Criteria:

1. Patients with hypertension, hyperglycemia, and hyperlipidemia caused by secondary metabolic syndrome (disease, drugs, surgery, etc.);
2. Patients with severe primary diseases such as heart, liver, kidney, lung, brain, endocrine, hematopoietic system in the past or at the time of enrollment;
3. Those who are confirmed to have acute coronary syndrome, malignant arrhythmia, and other serious heart diseases;
4. Patients with co-infection, malignant tumors or mental illness;
5. Patients with Cushing syndrome;
6. Patients with allergies or allergies to this drug;
7. Pregnant or breastfeeding women;
8. Those who have adjusted hypoglycemic, lipid-lowering, antihypertensive drugs or taking weight-loss drugs within 1 month before enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of changes in waist-to-hip ratio at 12 weeks | 12 weeks
  Measure and record the waist-to-hip ratio of the patient before and after treatment
Analysis of body mass index changes in 12 weeks | 12 weeks
  Measure and record the patient's BMI before and after treatment

SECONDARY OUTCOMES:
Improvement of the conversion score of phlegm-damp constitution judgment | 12 weeks
  To study the improvement of the conversion score of phlegm-damp constitution before and after treatment
Lipid Index | 4 weeks，8 weeks，12 weeks
  Investigate the changes in triglycerides, high-density lipoprotein cholesterol, cholesterol and low-density lipoprotein cholesterol during treatment
Fasting blood glucose index | 4 weeks，8 weeks，12 weeks
  Investigate changes in fasting blood glucose during treatment
2h blood glucose after meal | 4 weeks，8 weeks，12 weeks
  Investigate changes in 2h blood glucose after meal during treatment
HOMAA insulin resistance index | 12 weeks
  To investigate the changes of HOMAA insulin resistance index during treatment
Blood pressure index | 4 weeks，8 weeks，12 weeks
  Observe the changes in systolic and diastolic blood pressure during treatment
Inflammatory factors | 12 weeks
  Investigate the changes of hypersensitivity C-reactive protein and endotoxin during treatment

IPD SHARING:
Plan to Share IPD: Undecided